CLINICAL TRIAL: NCT03912064
Title: A Phase 1 Trial of CD25/Treg-depleted DLI Plus Ipilimumab for Myeloid Disease Relapse After Matched-HCT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-142; 5P01CA229092-05 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasms; Chronic Myelomonocytic Leukemia; Myelofibrosis
Keywords: Myelofibrosis; Chronic Myelomonocytic Leukemia; Myeloproliferative Neoplasms; Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Primary Myelofibrosis | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD25/Treg-depleted DLI + Ipilimumab (Experimental): * Ipilimumab is administered intravenously every 12 weeks
  * Patients will receive a defined dose of CD25hi Treg depleted DLI intravenously
  Interventions: Drug: Ipilimumab; Biological: CD25hi Treg depleted DLI

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab is an antibody that acts against CTLA-4
  Other Names: Yervoy
Biological: CD25hi Treg depleted DLI — Donor lymphocyte product

SUMMARY:
In this research study, our main goal for the ipilimumab portion of the study is to determine the highest dose of ipilimumab that can be given safely in several courses and to determine what side effects are seen in patients with Acute Myeloid Leukemia (AML), Myelodysplastic Syndromes (MDS), Myeloproliferative Neoplasms (MPN), Chronic Myelomonocytic Leukemia (CMML), or Myelofibrosis (MF).

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The U.S. Food and Drug Administration (FDA) has not approved ipilimumab for this specific disease but it has been approved for other uses. This drug has been used in other research studies and is now FDA-approved for the treatment of melanoma. Many people have also received ipilimumab on research studies for possible treatment of prostate cancer, lymphoma, kidney cancer, ovarian cancer and HIV infection. Information from those other research studies suggests that ipilimumab may help to treat the participant's cancer.

Ipilimumab is an antibody that acts against CTLA-4. An antibody is a common type of protein produced by the body that the immune system (a system that defends the body against potentially harmful particles) uses to find and destroy foreign molecules (particles not typically found in the body) such as bacteria and viruses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapse of AML, MDS or MPN (CMML or myelofibrosis or MDS/MPN with ≥5% blasts in the marrow).
* Relapse at ≥2 months after any 8/8 or better HLA-matched HCT
* Available original stem cell donor.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of Ipilimumab in participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky performance status ≥60, see Appendix A).
* Recipient donor T cell chimerism ≥20% within 4 weeks prior to cell infusion.
* <50% bone marrow involvement within 4 weeks prior to cell infusion.
* No systemic corticosteroid therapy for GVHD (≤5 mg of prednisone or equivalent doses of other systemic steroids for non-GVHD, non-autoimmune indications for at least 4 weeks prior to cell infusion).
* No other systemic medications/treatments (e.g. ECP) for GVHD for at least 4 weeks prior to cell infusion.
* Ability to understand and willingness to sign written informed consents.
* Adequate organ function as defined below:

  * Total bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * creatinine clearance: ≤1.5 x institutional ULN
  * O2 saturation: ≥90% on room air
  * LVEF >40%
* The effects of CD25/Treg-depleted DLI and Ipilimumab on the developing human fetus are unknown. For this reason and because immunomodulatory agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study or within 23 weeks after the last dose of study drug, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for at least 31 weeks after completion of Ipilimumab administration.
* Negative pregnancy test for females of childbearing potential only

Exclusion Criteria:

* Extramedullary relapse involving immuno-privileged sites (e.g. CNS, testes, eyes). Other sites of extramedullary relapse (e.g. leukemia cutis, granulocytic sarcoma) are acceptable.
* Participants who have had anti-tumor chemotherapy or other investigational agents within 4 weeks prior to cell infusion (6 weeks for nitrosoureas or mitomycin C), or immunotherapy within 8 weeks prior, or those who have not recovered from adverse events due to agents administered more than 4 weeks prior. Use of hydroxyurea to control counts within 4 weeks prior to cell infusion is permitted.
* Prior history of DLI
* Prior history of treatment with anti-CTLA-4 or anti-PD-1 pathway therapy, or CD137 agonist therapy.
* Prior history of severe (grade 3 or 4) acute GVHD, or ongoing active GVHD requiring systemic treatment.
* Organ transplant (allograft) recipient.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ipilimumab or other agents used in study.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis). Patients with Hashimoto's thyroiditis are eligible to go on study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the unknown teratogenic risk. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow- suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after HCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level: 0: 1 mg/kg of Ipilimumab and 3x10^7 CD3+ cells/kg of CD25/Treg-depleted DLI will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
- Dose Level: 1: 3 mg/kg of Ipilimumab and 3x10^7 CD3+ cells/kg of CD25/Treg-depleted DLI will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
- Dose Level: 2: 10 mg/kg of Ipilimumab and 3x10^7 CD3+ cells/kg of CD25/Treg-depleted DLI will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
Period: Overall Study
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Started | 18 | 6 | 1
Completed | 1 | 0 | 0
Not Completed | 17 | 6 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Adverse reaction to Ipilimumab | 2 | 0 | 1
Not completed — Progression/Relapse | 7 | 3 | 0
Not completed — Prolonged treatment delays | 3 | 2 | 0
Not completed — Prohibited concomitant treatments | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level: 0: 1 mg/kg of Ipilimumab will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
- Dose Level: 1: 3 mg/kg of Ipilimumab will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
- Dose Level: 2: 10 mg/kg of Ipilimumab will be administered intravenously over 90 ± 10 minutes after the DLI product observation period is completed, and dosing will continue in 3-week intervals for 4 cycles, unless unacceptable toxicity or symptomatic disease progression occurs.
- Total: Total of all reporting groups
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2 | Total
Number analyzed (Participants) | 18 | 6 | 1 | 25
Age, Continuous [Median (Full Range); unit: years] | 65 [25 to 72] | 57.5 [20 to 77] | 68 [68 to 68] | 65 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 0 | 11
  Male | 11 | 2 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 6 | 1 | 22
  Black/African American | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Unknown/Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for DLI
Description: The primary objective of this study is to determine the safety (MTD) of CD25/Treg-depleted donor lymphocyte infusion (DLI) plus Ipilimumab in patients with myeloid relapse after matched-HCT. Participants will be evaluated for dose limiting toxicities (DLTs) at day 43. DLTs explained within section 5.4 of the protocol.
Time Frame: Day 43 (6 weeks)
Measure: Number; unit: cells/kg
Groups:
- CD25/Treg-depleted DLI: CD25hi Treg depleted DLI: Donor lymphocyte product -Patients will receive a defined dose of CD25hi Treg depleted DLI intravenously
  Ipilimumab: Ipilimumab is an antibody that acts against CTLA-4
  -Ipilimumab is administered intravenously every 12 weeks
Arm/Group | CD25/Treg-depleted DLI
Number analyzed (Participants) | 25
cells/kg | 30000000

2. Primary Outcome: Maximum Tolerated Dose (MTD) for Ipilimumab
Description: as for outcome 1
Time Frame: Day 43 (6 weeks)
Measure: Number; unit: mg/kg
Groups:
- Ipilimumab: Ipilimumab: Ipilimumab is an antibody that acts against CTLA-4 -Ipilimumab is administered intravenously every 12 weeks
  CD25hi Treg depleted DLI: Donor lymphocyte product
  -Patients will receive a defined dose of CD25hi Treg depleted DLI intravenously
Arm/Group | Ipilimumab
Number analyzed (Participants) | 25
mg/kg | 1

3. Secondary Outcome: Response Rate as Determined by Complete Remission (CR) and CR With Incomplete Count Recovery (CRi)
Description: Complete remission will be evaluated for each disease, along with duration of complete remission. AML morphological complete remission can be found in Appendix E (E.1.1.), and Relapse from CR/CRi is in E.1.3. MDS/MPN complete remission criteria is found in Appendix F (F.1.1), and criteria for relapse is found in F.1.5.
Time Frame: Day 43 (6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
Participants | 8 | 4 | 0

4. Secondary Outcome: Progression Free Survival
Description: Duration of time from start of treatment to time of objective disease progression or death, whichever comes first. AML progressive disease is defined in Appendix E (E.1.7.), and criteria for MDS/MPN is in Appendix F (F.1.4.).
Time Frame: Day 92 and Week 60
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
percentage of participants
  Day 92 | 50 [27 to 73] | 83 [53 to 100] | NA [NA to NA] — Progression event (died without progression) at day 65, Sample size too small to estimate the rate and CI
  Week 60 | 33 [11 to 55] | 17 [0 to 47] | NA [NA to NA] — Progression event (died without progression) at day 65, Sample size too small to estimate the rate and CI

5. Secondary Outcome: Overall Survival
Description: Duration of time from start of treatment to time of death.
Time Frame: Day 92 and Week 60
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
percentage of participants
  Day 92 | 89 [75 to 100] | 100 [NA to NA] — No death before 150 days, cannot estimate CI | NA [NA to NA] — Died at day 65, Sample size too small to estimate the rate and CI
  Week 60 | 61 [37 to 83] | 67 [29 to 100] | NA [NA to NA] — Died at day 65, Sample size too small to estimate the rate and CI

6. Secondary Outcome: Incidence of Acute GVHD Rates
Description: Incidence of aGVHD will be measured at the below time point, and grading severity of aGVHD will be standardized using the chart and information in Appendix C.
Time Frame: Day 92
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
Participants | 2 | 2 | 1

7. Secondary Outcome: Incidence of Chronic GVHD Rates
Description: Provider will assess study subject for severity of cGVHD per 2014 NIH consensus criteria at day 92.
Time Frame: Day 92
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
Participants | 7 | 1 | 0

8. Secondary Outcome: Severity of Acute GVHD Rates
Description: Severity of aGVHD will be measured at the below time point, and grading severity of aGVHD will be standardized using the chart and information in Appendix C per Harris et al, 2016 "GVHD Target Organ Staging", where 0 is no GVHD and 4 is severe. For the data table below: Grade I-IV reports any incidence of aGVHD, Grade II-IV reports the number of subjects who developed grade II, III, and IV aGVHD and Grade III-IV reports the number of subjects who developed Grade III and IV aGHVD.
  Grade 0: No stage 1-4 of any organ. Grade I: Stage 1-2 skin without liver, upper GI, or lower GI involvement. Grade II: Stage 3 rash and/or stage 1 liver and/or stage 1 upper GI and/or stage 1 lower GI.
  Grade III: Stage 2-3 liver and/or stage 2-3 lower GI, with stage 0-3 skin and/or stage 0-1 upper GI.
  Grade IV: Stage 4 skin, liver, or lower GI involvement, with stage 0-1 upper GI.
Time Frame: Day 92
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
Participants
  Grade I-IV aGVHD | 2 | 2 | 1
  Grade II-IV aGVHD | 0 | 1 | 0
  Grade III-IV aGVHD | 2 | 1 | 1

9. Secondary Outcome: Severity of Chronic GVHD Rates
Description: Provider will assess study subject for severity of cGVHD per 2014 NIH consensus criteria at day 92.
Time Frame: Day 92
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
Number analyzed (Participants) | 18 | 6 | 1
Participants
  Mild cGVHD | 2 | 1 | 0
  Moderate cGVHD | 3 | 0 | 0
  Severe cGVHD | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are reported from the initial dose of study treatment through to 90 days after the last dose of treatment.
Description: An adverse event (AE) is any undesirable sign, symptom or medical condition or experience that develops or worsens in severity after starting the first dose of study treatment or any procedure specified in the protocol, even if the event is not considered to be related to the study. Infection: CTCAE gr 3 or less. And immune-related events (e.g. diarrhea, pruritus, rash, endocrinopathies) that respond to corticosteroids and improve to grade 1 or less with steroids: CTCAE gr 3 or less
Arm/Group | Dose Level: 0 | Dose Level: 1 | Dose Level: 2
All-Cause Mortality (participants affected / at risk) | 7/18 | 2/6 | 1/1
Serious Adverse Events (participants affected / at risk) | 4/18 | 2/6 | 1/1
Other Adverse Events (participants affected / at risk) | 18/18 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level: 0 (N=18) | Dose Level: 1 (N=6) | Dose Level: 2 (N=1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — GI bleed
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level: 0 (N=18) | Dose Level: 1 (N=6) | Dose Level: 2 (N=1)
Anemia (Blood and lymphatic system disorders) | 10 | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 0 — peripheral blood blast cells
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0 | 0 — Diabetic ketoacidosis
Dry eye (Eye disorders) | 1 | 0 | 0
Floaters (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — oral ulceration
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 12 | 1 | 0
Fever (General disorders) | 2 | 0 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 7 | 1 | 0 — cGVHD
Bacteremia (Infections and infestations) | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 11 | 4 | 1
Alkaline phosphatase increased (Investigations) | 7 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 3 | 1
Blood bilirubin increased (Investigations) | 6 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 8 | 1 | 1
CPK increased (Investigations) | 2 | 0 | 0
Creatinine increased (Investigations) | 4 | 2 | 0
Lipase increased (Investigations) | 6 | 1 | 1
Neutrophil count decreased (Investigations) | 11 | 1 | 0
Platelet count decreased (Investigations) | 12 | 2 | 0
Serum amylase increased (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 11 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — melanoma to small area of left scapula
Ataxia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Dysphasia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 — Aphasia
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Uterine pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 2 | 2 | 1 — aGVHD
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — Enteritis
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 0 — Diabetic Ketoacidosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT03912064/Prot_SAP_000.pdf